CLINICAL TRIAL: NCT01614730
Title: User Evaluation Trial in Healthy Volunteers : Modified Neurotech Vital Device
Brief Title: User Evaluation in Healthy Volunteers to Verify no Pelvic Floor Contraction is Stimulated When the Modified Neurotech Vital Device is Used Compared to the Neurotech Vital Device
Acronym: BMR-12-1002
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bio-Medical Research, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: BMR-12-1002
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-06

CONDITIONS: Contraction of Pelvic Floor Muscle Using EMS
Keywords: EMS; Modified Device
MeSH Terms: interventions — Emergency Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Neurotech Vital Device (Sham Comparator): Checking to see no contraction is stimulated during treatment with the Modified Neurotech Device
  Interventions: Device: Modified Neurotech Vital Device
- Neurotech Vital Device (Active Comparator): Checking to see a contraction is stimulated during treatment of the Neurotech Vital Device
  Interventions: Device: Neurotech Vital Device

INTERVENTIONS:
Device: Modified Neurotech Vital Device — verify no contraction is stimulated in the Modified Neurotech Vital.
  Other Names: Modified Neurotech Vital Device, EMS
  Arms: Modified Neurotech Vital Device
Device: Neurotech Vital Device — Checking there is a contraction of the pelvic floor muscle when the treatment is administered with the Neurotech Vital Device
  Other Names: EMS, Neurotech Vital
  Arms: Neurotech Vital Device

SUMMARY:
This user evaluation study is to verify that the Modified Neurotech Vital Device does not stimulate the pelvic floor muscles compared with the Neurotech Vital Device.

DETAILED DESCRIPTION:
This user evaluation study is to verify that the Modified Neurotech Vital Device does not stimulate the pelvic floor muscles compared with the Neurotech Vital Device. Stimulation of the pelvic floor muscles will be assessed by using sonographic/real time ultrasound imaging/recording with displacement measurement using onscreen callipers on the sonogram unit to assess contractions.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following inclusion criteria will be included in the study.

* Subjects who are female and at least 18 years of age.
* Subjects who, in the opinion of the Investigator, are deemed healthy.
* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained.
* Subjects who are able to understand this study and are willing to complete all the study assessments.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from participation in the study.

  * Subjects who have an existing medical condition that would compromise their participation in the study.
  * Subjects who have a physical condition that would make them unable to perform the study procedures.
  * Subjects with a history of any respiratory condition including a chronic cough.
  * Subjects with a history of an underlying neurological condition.
  * Subjects with a history of low back pain involving the spinal nerve root.
  * Subjects with a blood clotting disorder or who are taking anti-coagulant medications.
  * Subjects who have previously had any uro-gynaecological related surgery excluding hysterectomy.
  * Subjects with a clinical diagnosis of prolapse greater than Stage 2.
  * Subjects who are pregnant or could be pregnant.
  * Subjects who are less than 6 months post-partum or who are lactating.
  * Subjects who have any intra-uterine devices or metal implants in the pelvic area, including hip and lumbar spine.
  * Subjects with pelvic pain or fibromyalgia or paravaginal defect.
  * Subjects with an active implanted medical device (ie pacemaker, pump etc).
  * Subjects with a history of heart disease or stroke.
  * Subjects with a known cancer.
  * Subjects with an injury or disability affecting any part of their body which will be in contact with the garment.
  * Subjects who are currently involved in any injury litigation claims.
  * Subjects who have been committed to an institution by virtue of an order issued either by the courts or by an authority.
  * Subjects who have participated in a clinical study in the last 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Using a sonographic/real time ultrasound imaging machine detect if a contraction is stimulated by the 5 minute treatment with the modified Neurotech Device and 5 minute treatment with the Neurotech Vital Device. | 5 minutes treatment with each device to measure if contraction occurrs on the ultrasound
  The primary endpoint of the study is to demonstrate that no volunteers elicit a contraction of the pelvic floor muscle with the Modified Neurotech Vital Device and that all the volunteers elicit a contraction of the pelvic floor muscle with the Neurotech Vital Device. Contraction of the pelvic floor muscles will be assessed by using sonographic/real time ultrasound imaging/recording (mean of three measurements of pelvic floor displacement achieved during maximum threshold intensity electrical stimulation).

SECONDARY OUTCOMES:
Healthy Volunteers feedback questionnaires | after 5 minutes of treatment
  The secondary objective of this user evaluation study is to verify that the Modified Neurotech Vital Device is perceived by the volunteers as a valid treatment option. The Modified Neurotech Vital Device will be considered an acceptable treatment option in relation to stimulation sensation if 70% yes/not sure responses are obtained to the question 'given what you have been told about this treatment, do you believe it could be effective?'.